CLINICAL TRIAL: NCT03988751
Title: Real-time Location System Feasibility Study Part 2
Brief Title: Real-time Location System Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00039439
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Surgery; Mobility
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Ambulation (Active Comparator): The total distance will be 40 meters. Study team members will walk, support, and coach the subject to walk as slow as he/she wants
  Interventions: Behavioral: Ambulation
- Interval Ambulation (Active Comparator): The subject will walk a total distance of 40 meters. This distance will be divided into four intervals of 10 meters to equal the same measured distance as the continuous group. The subject will receive two minutes of rest between each interval and will be supported and coached to walk as fast as they can.
  Interventions: Behavioral: Ambulation

INTERVENTIONS:
Behavioral: Ambulation — Variation in ambulatory intensity.

SUMMARY:
The proposed study will investigate the feasibility of using the Wake Forest Real-time Location System (RTLS) in monitoring patient movement during their in-hospital postoperative recovery. The study will involve patients who have undergone surgery requiring inpatient admission to the surgical ward. Actual patient movement will be monitored during their postoperative recovery and compared with data recorded by the Wake Forest location system.

In this small pilot study, a subgroup of participants will be randomized to two cohorts, continuous walking and interval walking. Tolerability of the varied walking intensity will be measured.

ELIGIBILITY:
Inclusion criteria

* Male or female patients between the ages of 18 and 90.
* Admitted to the Surgical Ward.
* Recovering from surgery.
* Ability to understand and the willingness to sign an Institutional Review Board-approved informed consent document.
* Ability to understand and complete the study survey instruments in English.

Exclusion criteria

* Non-surgical patient.
* Emergency surgical procedure.
* Anticipated discharge less than 24 hour.
* Unable to ambulate or ambulation not permitted by treating provider.
* Unable to understand and complete the study survey instruments in English.
* Post-operative complications that in the opinion of the study investigator would impair the ability of the patient to adhere to the study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2022-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Ambulation: The total distance will be 40 meters. Study team members will walk, support, and coach the subject to walk as slow as he/she wants. Ambulation speed and duration per patient.
Period: Overall Study
Arm/Group | Continuous Ambulation | Interval Ambulation
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Continuous Ambulation: The subject will walk a total distance of 40 meters. Study team members will walk, support, and coach the subject to walk as slow as he/she wants.
- Total: Total of all reporting groups
Arm/Group | Continuous Ambulation | Interval Ambulation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [63 to 68] | 64 [51 to 65] | 64 [58 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Characterize Number of Participants Who Tolerate Continuous vs Interval 40m Walk.
Description: Characterize number of participants who tolerate continuous vs interval 40m walk by evaluation of adverse events and change in vital signs.
Time Frame: 1 day
Population: Number of participants who completed 40 meter ambulation without adverse event or significant change in vital signs
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Ambulation | Interval Ambulation
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Continuous Ambulation | Interval Ambulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03988751/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03988751/ICF_001.pdf